CLINICAL TRIAL: NCT00946881
Title: A Prospective, Multicenter Phase I/II Safety and Tolerability Study of Unilateral Vascular-Targeted Photodynamic Therapy Using WST11 in Patients With Localized Prostate Cancer
Brief Title: Safety and Tolerability Study Using WST11 In Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Steba Biotech S.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN901 PCM202
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
Keywords: Prostatic disease; genital neoplasm, male; Urogenital neoplasm; Genital disease; male; Male urogenital disease; Neoplasms; Neoplasm by site; prostatic neoplasm; Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases; Genital Neoplasms, Male; Urogenital Neoplasms; Genital Diseases; Male Urogenital Diseases; Neoplasms; Neoplasms by Site; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WST11 (TOOKAD® Soluble) (Experimental): WST11-mediated-VTP The WST11-mediated VTP procedure will consist of a single, 10 min, IV administration of WST11 at doses of either 2mg/kg, 4 mg/kg or 6 mg/kg, followed by light activation delivered through one or more transperineal interstitial optical fibers using 753 nm laser light at escalating fixed energy doses
  Interventions: Drug: WST 11 -mediated -VTP

INTERVENTIONS:
Drug: WST 11 -mediated -VTP — The WST11-mediated VTP procedure will consist of a single, 10 min, IV administration of WST11 at doses of either 2mg/kg, 4 mg/kg or 6 mg/kg, followed by light activation delivered through one or more transperineal interstitial optical fibers for 20 minutes using 753 nm laser light at escalating fixed energy doses of 200 J/cm and 300 J/cm, by escalating power at each energy to 167 mW/cm and 250 mW/cm, respectively. A brachytherapy-like template is used for the placement of the optical fiber(s) that are positioned in the prostate areas of interest under trans-rectal ultrasound image guidance.
  Other Names: TOOKAD Soluble

SUMMARY:
The aim of this study is to determine the optimal treatment conditions (WST11 dose and light energy dose) to achieve ablation in one lobe of the prostate and to evaluate the safety and quality of life of WST11 medicated Vascular-Targeted Photodynamic therapy (VTP) in men with localized prostate cancer.

DETAILED DESCRIPTION:
This study is designed as a multicenter, phase I/II, prospective, open-labeled, single intravenous (IV) dose, clinical trial in patients with localized prostate cancer.

The study population will be men who have been offered curative therapy (radical prostatectomy; cryotherapy; brachytherapy; External Beam RadioTherapy (EBRT), and refused. Patients must have already had a previous biopsy showing a histologically proven carcinoma of the prostate. The identification and the location of the tumor will be done using both dynamic contrast Magnetic resonance Imaging (MRI) and biopsy.

Only unilateral treatment with WST11-medicated VTP will be performed during the study. Treatment will consist of a single, 10 minute, IV administration of WST11 at doses of 2mg/kg, 4 mg/kg or 6 mg/kg, followed by either light activation delivered through transperineal interstitial optical fibers for 20 minutes using 753 nm laser light at escalating fixed energy doses of 200 J/cm or 300 J/cm by escalating power at each energy to 167 mW/cm or 250 mW/cm respectively. A brachytherapy-like template is used for the placement of the transparent implant catheters which are positioned in the prostate under transrectal ultrasound image guidance. The illumination fiber(s) are then inserted into the implant catheters.

If the safety profile for a given WST11 and light dose is acceptable, additional patients may be treated with multiple fibers at that WST11 treatment dose.

For cases where the Month 6 biopsy is positive, the patient will be offered the opportunity to be retreated with WST11

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosed with localized, prostate cancer and who have been offered curative therapy (radical prostatectomy; cryotherapy; brachytherapy; External Beam RadioTherapy (EBRT), and refused
* Localized prostate cancer stage T1C up to T2A based on biopsy performed at least 6 weeks prior to enrollment
* Gleason score ≤ 3+3 with ≤50% of sampled cores positive, and each positive core having a tumour length of ≤5 mm
* Prostate Specific Antigen (PSA) < 10 ng/mL
* No prior treatment for prostate cancer
* Signed Informed Consent Form

Exclusion Criteria:

* Any condition or history of illness or surgery that, in the opinion of the investigator and/or the Sponsor, might confound the results of the study or pose additional risks to the patient.
* All patients whose current pre-operative cardiac evaluation does not show their fitness for a procedure requiring general anesthesia;
* Patients with a prior history of viral or alcoholic hepatitis, and other patients felt to be at risk for hepatotoxicity including concomitant use of potentially hepatotoxic medications or dietary supplements;
* Patients with a history of inflammatory bowel disease or other factors which may increase the risk of fistula formation;
* Patients who have received any hormonal manipulation (excluding 5-alpha reductase inhibitors) or androgen supplements within the previous 6 months;
* Patients previously treated by radiation therapy (external therapy or brachytherapy) or chemotherapy or any therapy for prostate cancer;
* Patients who have received or are receiving chemotherapy for prostate carcinoma or other significant cancer;
* Patients who have undergone previous TURP (trans-urethral resection of the prostate);
* Patients with a history of urethral stricture disease
* Patients with a history of acute urinary retention
* Patients who are currently (within 10 days before the treatment procedure) receiving any medications having potential photosensitizing effects (e.g. tetracyclines, sulfonamides, phenothiazines, sulfonylurea hypoglycemic agents, thiazide diuretics and griseofulvin)
* Patients who are currently receiving anticoagulant drugs (within 10 days before the treatment procedure) (e.g.: coumadin, warfarin)
* Patient who stopped long term treatment of acetylsalicylic acid (aspirin) or other anti platelets agents within 10 days prior to the treatment procedure;
* Patient suspected of Disseminated Intravascular Coagulation (DIC) as defined by the presence of three out of the five following criteria: platelets decrease, increase of PT, increase of aPTT, fibrinogen decrease, D-Dimer increase; from the normal laboratory ranges;
* Patient with a history of vasculitis or collagen vascular disease;
* History of non compliance with medical therapy and medical recommendations or an unwillingness or inability to complete patient self-administered questionnaires;
* Participation in a clinical study or receipt of an investigational treatment within the past 3 months;
* A history of porphyria;
* A history of sun hypersensitivity or photosensitive dermatitis;
* Renal disorders (blood creatinine > 1.5 x ULN) or known post mictional residue > 150cc
* Hepatic disorders (transaminases > ULN, bilirubin > ULN, GGT > ULN). In case of slight abnormalities, another exam could be performed. If the results are within normal ranges, then the patient can be included;
* Hematological disorders (white cells < 2500/mm3, neutrophils < 1500/mm3, platelets, < 140.000/mm3, Hb ≤ 10 g/dL);
* Patients with contra-indication to MRI (such as pace maker, metal prosthesis, etc.).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Taneja, Professor, Principal Investigator — Department of Urology, New York University Cancer Institute
Locations (5):
- United States (5):
  - UCLA - Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Midtown Urology & Midtown Urology Surgical Center, Atlanta, Georgia
  - Washington University School of Medicine- Barnes-Jewish Hospital, St Louis, Missouri
  - NYU Urology Associates, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
The data are available in case report form for each patient

REFERENCES:
- [Result] Taneja SS, Bennett J, Coleman J, Grubb R, Andriole G, Reiter RE, Marks L, Azzouzi AR, Emberton M. Final Results of a Phase I/II Multicenter Trial of WST11 Vascular Targeted Photodynamic Therapy for Hemi-Ablation of the Prostate in Men with Unilateral Low Risk Prostate Cancer Performed in the United States. J Urol. 2016 Oct;196(4):1096-104. doi: 10.1016/j.juro.2016.05.113. Epub 2016 Jun 9. PMID 27291652
- [Derived] Azzouzi AR, Barret E, Bennet J, Moore C, Taneja S, Muir G, Villers A, Coleman J, Allen C, Scherz A, Emberton M. TOOKAD(R) Soluble focal therapy: pooled analysis of three phase II studies assessing the minimally invasive ablation of localized prostate cancer. World J Urol. 2015 Jul;33(7):945-53. doi: 10.1007/s00345-015-1505-8. Epub 2015 Feb 25. PMID 25712310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty patients were included in the study by five different centers in the US. All 30 patients received the entire VTP procedure (first treatment phase).
  Two of them discontinued the study prior to Month 12. Eight patients who had positive biopsies at Month 6 entered in the retreatment phase. Only 7 of them actually received retreatment.
Groups:
- WST 11(TOOKAD® Soluble): WST 11-mediated-VTP
  WST 11 -mediated -VTP: The WST11-mediated VTP procedure will consist of a single, 10 min, IV administration of WST11 at doses of either 2mg/kg, 4 mg/kg or 6 mg/kg, followed by light activation delivered through one or more transperineal interstitial optical fibers for 20 minutes using 753 nm laser light at escalating fixed energy doses of 200 J/cm and 300 J/cm, by escalating power at each energy to 167 mW/cm and 250 mW/cm, respectively. A brachytherapy-like template is used for the placement of the optical fiber(s) that are positioned in the prostate areas of interest under trans-rectal ultrasound image guidance.
Period: First Treatment
Arm/Group | WST 11(TOOKAD® Soluble)
Started | 30
Completed | 28
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Patient relocated to another state | 1
Period: Retreatment
Arm/Group | WST 11(TOOKAD® Soluble)
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All 30 patients were males suffering from low risk prostate cancer.
Arm/Group | WST 11(TOOKAD® Soluble)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Prostate Biopsy
Description: Arm/Group Title:
  WST 11(TOOKAD® Soluble) Arm/Group Description To define the study drug and light dosage combination to achieve negative biopsy in the treated lobe
Time Frame: Month 6
Measure: Number; unit: participants
Groups:
- 2 mg/Kg-200 J/cm: Number of patients with positives or négatives biopsies at the dose 2mg/Kg-200J/cm
- 2 mg/Kg-300 J/cm: Number of patients with positives or négatives biopsies at the dose 2mg/Kg-300J/cm
- 4 mg/Kg-200 J/cm: Number of patients with positives or négatives biopsies at the dose 4mg/Kg-200J/cm
- All Doses/Energies: Number of patients with positives or négatives biopsies at all doses/energies
Arm/Group | 2 mg/Kg-200 J/cm | 2 mg/Kg-300 J/cm | 4 mg/Kg-200 J/cm | All Doses/Energies
Number analyzed (Participants) | 3 | 6 | 21 | 30
participants
  Positive | 0 | 3 | 8 | 11
  Negative | 3 | 3 | 13 | 19

2. Primary Outcome: Prostate Biopsies
Description: Number of patients who had a negative biopsy at Month-6
Time Frame: Month-6
Measure: Count of Participants; unit: Participants
Groups:
- 2 mg/Kg-200 J/cm: Number of patients with negative biopsies at the dose 2mg/Kg-200J/cm
- 2 mg/Kg-300 J/cm: Number of patients with negative biopsies at the dose 2mg/Kg-300J/cm
- 4 mg/Kg-200 J/cm: Number of patients with negative biopsies at the dose 4mg/Kg-200J/cm
- All Doses/Energies: Number of patients with negative biopsies at all doses/energies
Arm/Group | 2 mg/Kg-200 J/cm | 2 mg/Kg-300 J/cm | 4 mg/Kg-200 J/cm | All Doses/Energies
Number analyzed (Participants) | 3 | 6 | 21 | 30
Participants | 3 | 3 | 13 | 19

3. Secondary Outcome: Pharmacokinetic Parameters-Cmax
Description: For each dose group, several pharmacokinetics parameters have been calculated.
Time Frame: T0, 5 min,10 min, 4 h, 8 h, post dose
Population: Out of 30 patients treated in the study, 29 patients had pharmacokinetic data available.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 2 mg/kg: Patients treated at the dose of 2 mg/kg of TOOKAD soluble, regardless of the dose of light, are analysed in this group.
- 4 mg/kg: Patients treated at the dose of 4 mg/kg of TOOKAD soluble, regardless of the dose of light, are analysed in this group.
Arm/Group | 2 mg/kg | 4 mg/kg
Number analyzed (Participants) | 9 | 20
ng/mL | 30883.83 (11583.07) | 57102.87 (14849.50)

4. Secondary Outcome: Percentage of Prostatic Necrosis at Day 7 as Observed on the 7-Day MRI
Description: The adjusted prostate necrosis percentage was defined as follows:
  The Day 7 necrosis percentage is the proportion, expressed in %, of Day 7 prostate necrosis volume by planimetry in the treated lobe compared with half the prostate volume by planimetry, considering the average between the baseline volume and Day 7 volume;
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: percentage of prostatic necrosis
Groups:
- 2 mg/Kg-200 J/cm: To evaluate the volume of necrosis observed on the 7-Day MRI in patients treated with 2 mg/kg-200J/cm
- 2 mg/Kg-300 J/cm: To evaluate the volume of necrosis observed on the 7-Day MRI in patients treated with 2 mg/kg-300J/cm
- 4 mg/Kg-200 J/cm: To evaluate the volume of necrosis observed on the 7-Day MRI in patients treated with 4 mg/kg-200J/cm
- All Doses/Energies: To evaluate the volume of necrosis observed on the 7-Day MRI in patients treated with all doses/energies
Arm/Group | 2 mg/Kg-200 J/cm | 2 mg/Kg-300 J/cm | 4 mg/Kg-200 J/cm | All Doses/Energies
Number analyzed (Participants) | 3 | 6 | 21 | 30
percentage of prostatic necrosis | 46.9 (41.6) | 13.8 (16.3) | 61.1 (25.3) | 52.3 (31.9)

5. Secondary Outcome: International Index of Erectile Functions (IIEF) Results
Description: The International Index of Erectile Functions questionnaire is 15 questions patients auto questionnaire. The results presented are those of the erectile function domain which comprise 6 questions. Possible scores range is 1 to 30 . Best score is 30, worst score is 1.
Time Frame: Month 1-Month 3- Month 6- Month 12
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 2 mg/Kg-200 J/cm: To assess the QoL-IIEF in patients treated with the dose 2mg/Kg-200J/cm
- 2 mg/Kg-300 J/cm: To assess the QoL-IIEF in patients treated with the dose 2mg/Kg-300J/cm
- 4 mg/Kg-200 J/cm: To assess the QoL-IIEF in patients treated with the dose 4mg/Kg-200J/cm
- All Doses/Energies: To assess the QoL-IIEF in patients treated with all doses/energies
Arm/Group | 2 mg/Kg-200 J/cm | 2 mg/Kg-300 J/cm | 4 mg/Kg-200 J/cm | All Doses/Energies
Number analyzed (Participants) | 3 | 6 | 21 | 30
units on a scale
  Baseline | 21.33 (4.73) | 13.17 (8.70) | 18.80 (7.88) | 17.90 (7.99)
  Month 1 | 14.33 (10.97) | 14.00 (8.92) | 13.65 (8.98) | 13.79 (8.80)
  Month 3 | 19.33 (4.04) | 14.17 (10.26) | 14.84 (7.91) | 15.18 (8.04)
  Month 6 | 19.33 (1.53) | 15.00 (9.47) | 15.29 (7.46) | 15.63 (7.46)
  Month 12 | 21.67 (2.52) | 6.25 (10.50) | 15.29 (8.48) | 14.48 (9.26)

6. Secondary Outcome: International Prostate Symptom Score (IPSS) Results
Description: The International Prostate Symptom Score (IPSS) is a 7 questions patients auto-questionnaire about urinary symptoms. the possible scores range are 0 to 35 . Best score is 0 worst score is 35
Time Frame: Month 1, Month 3 , Month 6 , Month 12
Population: IPSS results
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 2 mg/Kg-200 J/cm: To assess the QoL-IPSS in patients treated with the dose 2mg/Kg-200J/cm
- 2 mg/Kg-300 J/cm: To assess the QoL-IPSS in patients treated with the dose 2mg/Kg-300J/cm
- 4 mg/Kg-200 J/cm: To assess the QoL-IPSS in patients treated with the dose 4mg/Kg-200J/cm
- All Doses/Energies: To assess the QoL-IPSS in patients treated with all doses/energies
Arm/Group | 2 mg/Kg-200 J/cm | 2 mg/Kg-300 J/cm | 4 mg/Kg-200 J/cm | All Doses/Energies
Number analyzed (Participants) | 3 | 6 | 21 | 30
units on a scale
  Baseline | 10.67 (8.02) | 11.67 (7.31) | 8.65 (6.82) | 9.48 (6.88)
  Month 1 | 9.67 (9.87) | 11.00 (6.00) | 10.62 (6.34) | 10.60 (6.38)
  Month 3 | 4.67 (5.69) | 8.83 (4.83) | 8.00 (5.36) | 7.83 (5.22)
  Month 6 | 9.67 (8.62) | 8.50 (4.23) | 6.71 (4.80) | 7.37 (5.02)
  Month 12 | 7.33 (4.04) | 15.5 (8.89) | 7.93 (4.50) | 9.29 (6.02)

7. Secondary Outcome: Pharmacokinetic Parameters-Tmax
Description: For each dose group, several pharmacokinetics parameters have been calculated.
Time Frame: T0, 5 min,10 min, 4 h, 8 h, post dose
Population: Out of 30 patients treated in the study, 29 patients had pharmacokinetic data available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 2 mg/kg | 4 mg/kg
Number analyzed (Participants) | 9 | 20
hours | 0.43 (0.61) | 0.25 (0.22)

8. Secondary Outcome: Pharmacokinetic Parameters -T1/2
Description: For each dose group, several pharmacokinetics parameters have been calculated.
Time Frame: T0, 5 min,10 min, 4 h, 8 h, post dose
Population: Out of 30 patients treated in the study, 29 patients had pharmacokinetic data available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 2 mg/kg | 4 mg/kg
Number analyzed (Participants) | 9 | 20
hours | 1.25 (0.90) | 1.69 (1.11)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- WST 11(TOOKAD® Soluble): WST 11-mediated-VTP The WST11-mediated VTP procedure will consist of a single, 10 min, IV administration of WST11 at doses of either 2mg/kg, 4 mg/kg or 6 mg/kg, followed by light activation delivered through one or more transperineal interstitial optical fibers using 753 nm laser light at escalating fixed energy doses
  WST 11 -mediated -VTP: The WST11-mediated VTP procedure will consist of a single, 10 min, IV administration of WST11 at doses of either 2mg/kg, 4 mg/kg or 6 mg/kg, followed by light activation delivered through one or more transperineal interstitial optical fibers for 20 minutes using 753 nm laser light at escalating fixed energy doses of 200 J/cm and 300 J/cm, by escalating power at each energy to 167 mW/cm and 250 mW/cm, respectively. A brachytherapy-like template is used for the placement of the optical fiber(s) that are positioned in the prostate areas of interest under trans-rectal ultrasound image guidance.
Arm/Group | WST 11(TOOKAD® Soluble)
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 25/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WST 11(TOOKAD® Soluble) (N=30)
Gastrointestinal disorder (Gastrointestinal disorders) | 9 (10)
General disorders (General disorders) | 5 (5)
Injury, poisoning (Injury, poisoning and procedural complications) | 3 (3)
Investigations (Investigations) | 9 (12)
Musculoskeletal disorders (Musculoskeletal and connective tissue disorders) | 5 (6)
Nervous system disorders (Nervous system disorders) | 2 (2)
Renal and urinary disorders (Renal and urinary disorders) | 19 (45)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 16 (25)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin disorders (Skin and subcutaneous tissue disorders) | 5 (5)
Vascular disorders (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less